CLINICAL TRIAL: NCT05401981
Title: Disjunction Between Patient Narrative and Formulaic Thinking in the Doctor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Deemed not feasible.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, David Ring, MD, PhD Associate Dean for Comprehensive Care, Professor of Surgery and Psychiatry, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-01-0115
Record Dates: First submitted 2022-05-11; First posted 2022-06-02 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Diseases
Keywords: Orthopedics
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will randomly be assigned to 2 groups of intervention (The clinician receives the check list) and control (The clinician doesn't receive a checklist). After the visit patients will answer to questionnaires .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Clinician not given any cards about the patient's story.
- Story checklist (Experimental): Clinician given a card with talking points in the form of a checklist about the patient's story.
  Interventions: Other: Story checklist

INTERVENTIONS:
Other: Story checklist — The story checklist consists of a couple of questions that gives the physician something to keep in mind while visiting the patients.
  Arms: Story checklist

SUMMARY:
This study is seeking whether giving or not giving a clinician a card with talking points in the form of a checklist about the patient's story affects the patients care experience or not

DETAILED DESCRIPTION:
During an office visit, the clinician and the patient engage in dialogue and begin a relationship. This traditionally starts with the patient telling their story, which conveys why they decided to seek care. This study will determine the influence of a checklist specifically about the patient's narrative. The checklist will be used during the interview portion of the visit, to remind the clinician to stay curious about the person before them, their experience of the illness, and their explanatory model, and to help ensure that empathic opportunities are not missed.

ELIGIBILITY:
Inclusion Criteria:

* New patients
* Orthopedic visit

Exclusion Criteria:

* Languages other than English or Spanish.
* Cognitive dysfunction precluding completion of questionnaires.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient Experience Measure questions | through study completion, an average of 6 months
  Questionnaire assessing patient's experience

SECONDARY OUTCOMES:
Perceived empathy (JSPPPE) | through study completion, an average of 6 months
  Patient perceived of physician empathy as measured by the JSPPPE;The scores range from 1 ("Strongly Disagree") to 7 ("Strongly Agree"), with the total score being between 5 and 35. Higher scores represent greater empathic perception about the physician.
Guttman | through study completion, an average of 6 months
  Patient Satisfaction as measured by the Guttman Scale, The total score is between 0 and 7, with higher scores indicating greater satisfaction.
Guttman CEQ | through study completion, an average of 6 months
  Communication Effectiveness Questionnaire; The total score is the sum of all item scores (9 to 63) with higher scores representing a greater degree of perceived communication effectiveness.
PROMIS PF CAT | through study completion, an average of 6 months
  Patient Physical Function is measure by the PROMIS PF CAT; Higher scores indicate better physical function, with a mean of 50 for the general US population
NRS pain intensity assessment | through study completion, an average of 6 months
  Numeric rating scale = 11 point ordinal scale, the higher score indicates the more pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — The University of Texas at Austin
Locations (5):
- United States (5):
  - Austin Regional Clinic, Austin, Texas
  - Texas Orthopedics, Austin, Texas
  - HTB Musculoskeletal Institute, Austin, Texas
  - Orthopedic Specialists of Austin, Austin, Texas
  - ATX Ortho, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided